CLINICAL TRIAL: NCT00328679
Title: Food-Specific IgE, IgG, IgG4, Skin Prick Testing and Atopy Patch Testing in Children/Adolescents With Functional Dyspepsia: A Pilot Study
Brief Title: Evaluation of Food Hypersensitivity in Children/Adolescents With Functional Dyspepsia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Nancy Neilan, MT (ASCP)/ Research Coordinator, Children's Mercy Hospitals and Clinics
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0604-068
Record Dates: First submitted 2006-05-18; First posted 2006-05-22 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Dyspepsia
Keywords: abdominal; stomach; dyspepsia; food allergy
MeSH Terms: conditions — Dyspepsia; Food Hypersensitivity | interventions — In Vitro Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: in vitro and in vivo allergy testing

INTERVENTIONS:
Device: in vitro and in vivo allergy testing — Patch Test: food to be tested is suspended in sterile saline, placed on the skin of the back using a Finn Chamber secured with surgical tape and left in place for 48 hours.

SUMMARY:
The main purpose of this study is to determine if standard and investigational tests used to help diagnose and treat food allergies can provide information that will be useful in determining the cause of dyspepsia and helpful in designing a treatment plan. The study will also determine if there is a connection between positive allergy tests and inflammation in the upper abdomen.

DETAILED DESCRIPTION:
Recurrent abdominal pain is the most common type of pain in school age children and young adolescents. Over 80% of these children have pain in the upper abdomen which is diagnosed as functional dyspepsia (FD). Many of these children are also found to have eosinophilic duodenitis (ED). ED is a type of inflammation in the lining of the gastrointestinal tract characterized by an increase in eosinophils. An increase in intestinal eosinophils is a finding also seen with food allergy upon exposure to the offending antigen. The presence of intestinal eosinophilia in ED would suggest an allergic mechanism may be involved in the generation of pain and other symptoms associated with ED. Endoscopy and biopsy are used to aid in the identification of ED, which often is followed by elimination diets and food challenges to identify the offending allergen. This approach is both invasive (due to endoscopy) and cumbersome (due to the complexity and restrictiveness of the elimination diet). The value of screening for food hypersensitivities in children with ED has not been well characterized despite the theoretical links between food hypersensitivities, gut inflammation, and symptoms of dyspepsia. The current study will determine if standard and investigational tests used to evaluate food hypersensitivity have the potential to be used as biomarkers to direct treatment of children with ED.

ELIGIBILITY:
Inclusion Criteria:

* Age of 8-17 years, inclusive
* Diagnosis of functional dyspepsia (FD) by physician based on Rome II criteria (patient group only)
* Undergoing endoscopy to evaluate FD following demonstration of a lack of clinical response to acid reduction therapy (patient group only)
* Informed permission/assent

Exclusion Criteria (patient goup):

* Previous testing for food-specific IgE, IgG, IgG4, skin prick or allergy patch tests within the past 12 months or any previous positive result(s) for food-specific IgE, IgG, IgG4, SPT or APT to milk, egg, soy, corn, peanut or wheat;
* Any use of steroids or leukotriene receptor antagonists within one month prior to the study
* Any use of antihistamines, antihistamine-like drugs or topical steroid within two weeks prior to the study
* Any chronic non-gastrointestinal illness requiring regular medical care

Exclusion Criteria (healthy control group)

* In addition to patient exclusion criteria as defined above
* Any current or chronic history within the previous 6 months of gastrointestinal symptoms including abdominal pain or discomfort, nausea, vomiting, bloating, diarrhea or constipation
* History of asthma or chronic respiratory symptoms
* History of allergic rhinitis or chronic sinusitis
* History of allergic reactions attributed to food

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
measure specific IgE, IgG total, IgG subclass 4, skin prick tests and atopy patch tests to milk, egg, soy, corn, peanut and wheat | 48 hrs and 72 hrs after patch placement

SECONDARY OUTCOMES:
Determine T-lymphocytes, eosinophils and mast cell densities on duodenal biopsy samples demonstrating eosinophilia | collected at time of biopsy, patient group only

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Neilan, MT (ASCP), Principal Investigator — The Children's Mercy Hospital and Clinics
Locations (1):
- The Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Neilan NA, Dowling PJ, Taylor DL, Ryan P, Schurman JV, Friesen CA. Useful biomarkers in pediatric eosinophilic duodenitis and their existence: a case-control, single-blind, observational pilot study. J Pediatr Gastroenterol Nutr. 2010 Apr;50(4):377-84. doi: 10.1097/MPG.0b013e3181c2c28a. PMID 20216101